CLINICAL TRIAL: NCT03101241
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study of CX-8998 for Essential Tremor
Brief Title: A Phase 2 RCT Study of CX-8998 for Essential Tremor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CX-8998-CLN2-001
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Results first posted 2021-10-22 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-10

CONDITIONS: Essential Tremor
Keywords: Essential Tremor; Movement Disorders; thalamocortical dysrhythmias
MeSH Terms: conditions — Essential Tremor; Movement Disorders

STUDY DESIGN:
Intervention Model Description: This is a double-blind, placebo-controlled, parallel-group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CX-8998 (Experimental)
  Interventions: Drug: CX-8998
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CX-8998 — T-type calcium channel blocker
  Arms: CX-8998
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
This is a multicenter, double-blind, placebo-controlled, parallel-group study consisting of a screening period of up to 4 weeks (with the exception of participants on primidone at baseline who will be allowed 6 weeks of screening to allow for safe discontinuation). Screening results from all patients meeting the eligibility requirements will be further assessed by the sponsor medical personnel for final approval of suitability for inclusion in the study. Randomized participants will enter a 4 week double-blind dose-titration treatment period, followed by a 1 week safety follow-up period following the last dose of study medication, and a scheduled follow-up safety telephone call one week later.

DETAILED DESCRIPTION:
This is a multicenter, double-blind, placebo-controlled, parallel-group study consisting of a screening period of up to 4 weeks (with the exception of participants on primidone at baseline who will be allowed 6 weeks of screening to allow for safe discontinuation). Screening results from all patients meeting the eligibility requirements will be further assessed by the sponsor medical personnel for final approval of suitability for inclusion in the study. Randomized participants will enter a 4 week double-blind dose-titration treatment period, followed by a 1 week safety follow-up period following the last dose of study medication, and a scheduled follow-up safety telephone call one week later.

Participants will be randomized to one of two treatment groups. Group A will receive titrating doses of CX-8998 up to 10 mg BID and Group B will receive placebo. Participant randomization will be stratified by presence or absence of a single concomitant anti-tremor medication and by site-type (sub-study vs non sub-study).

Tremor will be assessed via The Essential Tremor Rating Assessment Scale (TETRAS) and accelerometry. To reduce the potential for bias in the assessments of efficacy, all participants will be videotaped during the TETRAS performance scale testing according to a consistent script. The videotapes will be rated in a blinded manner by qualified, independent raters. A subset of participants will participate in a digital biomarker sub-study.

Participants will be screened up to 4 weeks prior to initiation of dosing. Participants taking primidone at screening who are otherwise deemed eligible for participation and are willing to discontinue primidone will be allowed an additional 2 weeks of screening (a total of 6 weeks) to ensure safe primidone discontinuation. At Baseline, participants will undergo safety and tremor assessments prior to dosing, will receive their first dose of study drug and will be monitored for safety for one hour following dosing. For one week participants will receive 4 mg (or matching placebo) twice daily. Participants will return to the clinic on Day 8 for safety monitoring and dose up-titration to 8 mg (or matching placebo) twice daily. At Day 15 (Week 3) participants will return to clinic for safety and efficacy assessments and final dose up-titration to 10 mg (or matching placebo) twice daily. The final efficacy visit will occur at Day 28 (Week 4). A final safety visit will occur at Day 35 (Week 5). Should participants experience intolerable adverse events (AEs) at 4 mg BID, 8 mg BID or 10 mg BID, the dose may be decreased at Day 8 or Day 15 to the next lowest dose one time (or 2 mg BID in the case of the 4 mg BID dose.

Randomized participants will have the opportunity to participate in an optional exploratory sub-study designed to assess the utility of digital assessment tools for tremor (sub-study addendum #1). Participants with Parkinson's disease tremor will be enrolled in a second exploratory sub-study (addendum #2).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form indicating that the subject has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential benefits, side effects, risks, and discomforts.
2. Men or non-pregnant, non-breastfeeding women 18 to 75 years-of-age who are able to read and understand English.
3. Diagnosis of definite or probable essential tremor (ET) as defined by the Tremor Investigational Group with involvement of the hands and arms without present causes of enhanced physiologic tremor (Deuschl et al.,1998).
4. Diagnosis of ET before the age of 65.
5. Tremor severity score of at least 2 in at least one upper extremity on at least one of the three maneuvers on the TETRAS scale.
6. Total TETRAS performance score of at least 15.
7. One concomitant anti-tremor medication (other than primidone) is allowed. Note: Primidone is NOT an allowed anti-tremor medication. If on primidone, subjects are allowed to extend their screening period by 2 weeks (for a total of 6 weeks) and discontinue primidone under the supervision of the investigator.
8. Subjects with reproductive capability including all males and women of child-bearing potential (WOCBP) must agree to practice continuous abstinence or adequate contraception methods (appropriate double barrier method or oral, patch, implant, or injectable contraception) from as soon as feasible during screening period until at least 30 days after the last dose.
9. Approval by the sponsor medical personnel as to final suitability for the study.

Exclusion Criteria:

1. Exposure to tremorigenic drugs or drug withdrawal states within the 30 days prior to the first planned dose of study drug.
2. Direct or indirect trauma to the nervous system within 3 months preceding the onset of tremor
3. History or clinical evidence of psychogenic tremor origin
4. Known history of other medical or neurological conditions that may cause or explain subject's tremor, including, but not limited to: a. Parkinson's disease b. dystonia c. cerebellar disease, other than essential tremor d. Traumatic Brain Injury e. alcohol abuse or withdrawal f. mercury poisoning g. hyperthyroidism h. pheochromocytoma i. head trauma or cerebrovascular disease within 3 months prior to the onset of essential tremor j. multiple sclerosis k. polyneuropathy l. family history of Fragile X syndrome
5. Prior MR-guided Focused Ultrasound or surgical intervention (e.g., deep brain stimulation, ablative thalamotomy or gamma knife thalamotomy).
6. Botulinum toxin injection in the 6 months prior to screening.
7. Currently using more than one anti-tremor medication.
8. Experiencing clinical benefit from and/or is not willing to discontinue primidone
9. Use of medication(s) in the past month that might produce tremor or interfere with the evaluation of tremor, such as, but not limited to: CNS-stimulants, lithium, amiodarone, metoclopramide, theophylline, and valproate
10. Inability to refrain from use of medication/substance(s) that might produce tremor or interfere with the evaluation of tremor on study visit days, such as but not limited to stimulant decongestants, beta-agonist bronchodilators, caffeine, alcohol and tobacco, based on Investigator assessment at baseline.
11. Positive urine drug screen.
12. Regular use of more than two units of alcohol per day.
13. Sporadic use of a benzodiazepine, sleep medication or anxiolytic to improve sleep performance. Stable use at a consistent dose is allowed as long as tremor persists against the background of regular medication use. Use on the evening prior to a study visit is prohibited.
14. Use of prescription or non-prescription drugs or other products (i.e. grapefruit juice) known to be strong inhibitors or inducers of CYP3A4 which cannot be discontinued 2 weeks prior to Day 1 of dosing and withheld throughout the study, including primidone.
15. Concurrent illnesses that would be a contraindication to trial participation, including, but not limited to: a. Severe arterial thromboembolic events (myocardial infarction, unstable angina pectoris, stroke) less than 6 months before screening b. NYHA Class III or IV congestive heart failure, ventricular arrhythmias or uncontrolled blood pressure c. Clinically significant ECG d. Known infection with HIV, hepatitis B, or hepatitis C, unless curative therapy completed for hepatitis C with negative PCR for HCV RNA e. Significant hepatic (AST/ALT > 2X upper limit of normal) or renal disease (creatinine clearance <39 mL/min) f. Significant psychiatric history including mood disorders and alcohol or substance abuse within the last year g. A current C-SSRS score of 4 or 5 at screening or history of suicide attempt at any time during the past year h. Clinically significant impaired balance or is considered at increased risk for falls i. Symptomatic orthostatic hypotension.
16. Treatment with an investigational agent within 30 days prior to the first dose of CX-8998 or planning to receive an investigational agent during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-07-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Tucson Neuroscience Research, Tucson, Arizona
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - University of California San Diego, La Jolla, California
  - Pacific Research Network, San Diego, California
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - University of South Florida, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Meridian Neurology Clinical Research, Savannah, Georgia
  - Northwestern Medical Group, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Boston University Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Quest Research Institute, Farmington Hills, Michigan
  - Henry Ford Hospital West Bloomfield, West Bloomfield, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - St. Louis Clinical Trials, St Louis, Missouri
  - Columbia University, New York, New York
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Midwest Clinical Research Center, Dayton, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - Houston Methodist Neurological Institute, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Papapetropoulos S, Lee MS, Boyer S, Newbold EJ. A Phase 2, Randomized, Double-Blind, Placebo-Controlled Trial of CX-8998, a Selective Modulator of the T-Type Calcium Channel in Inadequately Treated Moderate to Severe Essential Tremor: T-CALM Study Design and Methodology for Efficacy Endpoint and Digital Biomarker Selection. Front Neurol. 2019 Jun 11;10:597. doi: 10.3389/fneur.2019.00597. eCollection 2019. PMID 31244760

RESULTS

PARTICIPANT FLOW:
Groups:
- CX-8998: Participants were administered CX-8998 4 mg (2 capsules) BID in week 1, then 8 mg (4 capsules) BID in week 2, and then 10 mg (5 capsules) BID in weeks 3 and 4.
- Placebo: Participants were administered a Placebo comparator of 2 capsules BID in week 1, then 4 capsules BID in Week 2, and then 5 capsules BID in Weeks 3 and 4.
Period: Overall Study
Arm/Group | CX-8998 | Placebo
Started | 48 | 47
Completed | 37 | 42
Not Completed | 11 | 5
Not completed — Intercurrent condition necessitating discontinuation | 4 | 2
Not completed — Participant withdrew consent | 3 | 1
Not completed — Investigator decision that withdrawal was in best interest of participant | 2 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lack of efficacy/subject withdrew consent | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed using the Intent-to-Treat Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | CX-8998 | Placebo | Total
Number analyzed (Participants) | 48 | 47 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (9.6) | 63 (10.8) | 63 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 25 | 25 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 48 | 45 | 93
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 45 | 46 | 91
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Baseline and Day 28 on The Essential Tremor Rating Assessment Scale Performance Subscale (TETRAS-PS) Total Score
Description: The Essential Tremor Rating Assessment Scale Performance Subscale (TETRAS-PS) was used to assess the efficacy of CX-8998 in reducing essential tremor as scored by the independent video raters. TETRAS-PS quantifies tremor in the head, face, voice, limbs, and trunk. The overall subscale score ranges from a minimum of 0 to a maximum of 64. A lower score is indicative of improvement and a better outcome.
Time Frame: Baseline and Day 28 post-dose.
Population: TETRAS-PS was assessed using the Full Analysis Set. The number analyzed by Day 28 decreased due to participants that did not complete the study to that time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CX-8998 | Placebo
Number analyzed (Participants) | 39 | 44
score on a scale
  Baseline | 22.7 (6.44) | 22.8 (5.84)
  Day 28: number analyzed (Participants) | 38 | 43
  Day 28 | 21.1 (6.71) | 20.7 (7.96)

2. Primary Outcome: Change From Baseline to Day 28 on The Essential Tremor Rating Assessment Scale Performance Subscale (TETRAS-PS)
Description: The Essential Tremor Rating Assessment Scale Performance Subscale (TETRAS-PS) was used to assess the efficacy of CX-8998 in reducing essential tremor as scored by the independent video raters. TETRAS-PS quantifies tremor in the head, face, voice, limbs, and trunk. The overall subscale score ranges from a minimum of 0 to a maximum of 64. A decrease or negative change in the score is indicative of improvement in outcome.
Time Frame: Baseline up to Day 28 post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CX-8998 | Placebo
Number analyzed (Participants) | 38 | 43
score on a scale | -1.6 (4.36) | -2.0 (4.98)

3. Secondary Outcome: Baseline and Day 28 on The Essential Tremor Rating Assessment Scale Activities of Daily Living (TETRAS-ADL) Subscale Score
Description: TETRAS-ADL subscale assesses items such as eating and drinking, dressing and personal hygiene, carrying items, and finer motor skills. Each item is rated on a scale for 0 to 4 on which 0 = normal activity and 4 = severe abnormality. The sum of the individual scores provides an overall score, which ranges from a minimum of 0 to a maximum of 48. A lower score is indicative of improvement or a better outcome.
Time Frame: Baseline and Day 28 post-dose.
Population: TETRAS-ADL score was assessed using the Full Analysis Set. The number analyzed by Day 28 decreased due to participants that did not complete the study to that time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CX-8998 | Placebo
Number analyzed (Participants) | 39 | 44
score on a scale
  Baseline | 25.7 (6.00) | 26.0 (7.13)
  Day 28: number analyzed (Participants) | 37 | 42
  Day 28 | 21.5 (6.44) | 24.8 (9.19)

4. Secondary Outcome: Change From Baseline to Day 28 on The Essential Tremor Rating Assessment Scale Activities of Daily Living (TETRAS-ADL) Subscale Score
Description: TETRAS-ADL subscale assesses items such as eating and drinking, dressing and personal hygiene, carrying items, and finer motor skills. Each item is rated on a scale for 0 to 4 on which 0 = normal activity and 4 = severe abnormality. The sum of the individual scores provides an overall score, which ranges from a minimum of 0 to a maximum of 48. A decrease or negative change in score is indicative of improvement or a better outcome.
Time Frame: Baseline up to Day 28 post-dose.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CX-8998 | Placebo
Number analyzed (Participants) | 37 | 42
score on a scale | -4.2 (6.71) | -1.3 (6.35)

5. Secondary Outcome: Baseline and Day 28 in the Kinesia ONE Score
Description: Kinesia ONE was developed to provide a quantitative measurement of motor symptoms in individuals with Parkinson's disease. Scores are presented as the sum of the scores of the left and right hands. A total of 4 tasks were performed on the left side and then on the right side to assess resting, postural, kinetic, and lateral wing beating tremor. Values for each test range from 0 (no tremor) to 4 (severe tremor). The total overall score is the sum of all individual items and ranges from a minimum of 0 to a maximum of 32. A lower score is indicative of improvement or a better outcome.
Time Frame: Baseline and Day 28 post-dose.
Population: Kinesia ONE score was assessed using the Full Analysis Set. The number analyzed by Day 28 decreased due to participants that did not complete the study to that time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CX-8998 | Placebo
Number analyzed (Participants) | 39 | 44
score on a scale
  Baseline | 10.6 (4.33) | 12.0 (5.35)
  Day 28: number analyzed (Participants) | 37 | 41
  Day 28 | 9.3 (4.28) | 10.4 (4.84)

6. Secondary Outcome: Change From Baseline to Day 28 in the Kinesia ONE Score
Description: Kinesia ONE was developed to provide a quantitative measurement of motor symptoms in individuals with Parkinson's disease. Scores are presented as the sum of the scores of the left and right hands. A total of 4 tasks were performed on the left side and then on the right side to assess resting, postural, kinetic, and lateral wing beating tremor. Values for each test range from 0 (no tremor) to 4 (severe tremor). The total overall score is the sum of all individual items and ranges from a minimum of 0 to a maximum of 32. A decrease or negative change in score is indicative of improvement or a better outcome.
Time Frame: Baseline up to Day 28 post-dose.
Population: Change from baseline to Day 28 in the Kinesia ONE Score was assessed using the Full Analysis Set. The number analyzed by Day 28 decreased due to participants that did not complete the study to that time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CX-8998 | Placebo
Number analyzed (Participants) | 37 | 41
score on a scale | -1.4 (3.35) | -1.8 (3.00)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time the informed consent form was signed through the follow-up telephone call on Day 56. AEs were followed until resolution or until the symptoms or values returned to normal or acceptable limits, whichever was earlier.
Description: Treatment-emergent adverse events (TEAEs) are adverse events (AEs) that occur after the initiation of the study drug through 30 days after the last dose or a pretreatment event that worsens in intensity during the same period.
Arm/Group | CX-8998 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/47
Serious Adverse Events (participants affected / at risk) | 1/48 | 0/47
Other Adverse Events (participants affected / at risk) | 28/48 | 19/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CX-8998 (N=48) | Placebo (N=47)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CX-8998 (N=48) | Placebo (N=47)
Dizziness (Nervous system disorders) | 10 | 3
Headache (Nervous system disorders) | 4 | 2
Disturbance in attention (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 2 | 1
Somnolence (Nervous system disorders) | 1 | 2
Hypoaethesia (Nervous system disorders) | 0 | 2
Euphoric mood (Psychiatric disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 3 | 0
Abnormal dreams (Psychiatric disorders) | 2 | 1
Hallucination (Psychiatric disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 1
Tinnitus (Ear and labyrinth disorders) | 2 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-04-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT03101241/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT03101241/SAP_001.pdf